CLINICAL TRIAL: NCT06820099
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Phase II Clinical Study Evaluating the Efficacy and Safety of HRS-7535 in Subjects With Heart Failure, Mild Reduction/Preservation of Ejection Fraction, and Obesity
Brief Title: Study on the Efficacy and Safety of HRS-7535 in Patients With Mild Decrease in Ejection Fraction/Preserved Ejection Fraction Heart Failure and Obesity
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shandong Suncadia Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HRS-7535-206
Record Dates: First submitted 2025-02-06; First posted 2025-02-11 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-02

CONDITIONS: Adults With Heart Failure, Mild Decrease in Ejection Fraction/Preserved Ejection Fraction, and Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group A (Experimental)
  Interventions: Drug: HRS-7535 tablet
- Treatment group B (Placebo Comparator)
  Interventions: Drug: HRS-7535 tablet placebo

INTERVENTIONS:
Drug: HRS-7535 tablet — HRS-7535 tablet.
  Arms: Treatment group A
Drug: HRS-7535 tablet placebo — HRS-7535 tablet placebo.
  Arms: Treatment group B

SUMMARY:
This is a multicenter, randomized, double-blind, placebo-controlled, parallel design phase II clinical trial, including a screening period of up to 2 weeks, a 36-weeks' treatment period, and a 1-week safety follow-up visit period.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, on the day of signing the informed consent form, aged between 18 and 80 years old;
2. Diagnosed with chronic heart failure for at least 1 months before screening, and diagnosed with heart failure with preserved ejection fraction according to the National Heart Failure Guidelines 2023 during the screening period;
3. Screening period and day 1 randomization before New York Heart Association (NYHA) functional classification II-IV;
4. During the screening period and on the first day before randomization, the body mass index (BMI) was ≥ 28 kg/m2;
5. Self reported having controlled diet and exercise for 3 months or more before screening, and having a weight change of no more than 5kg within the first 3 months of screening and randomization
6. During the screening period and on the first day of randomization, the total clinical score (KCCQ-CSS) of the Kansas City Cardiomyopathy Questionnaire should be ≤ 80 points;
7. Visit 1 and Visit 2 each undergo a 6MWT, both of which must be ≥ 100 meters and ≤ 425 meters;
8. Prior to screening, the stable dose of medication for underlying diseases (excluding oral diuretics) should be ≥ 4 weeks;
9. Capable and willing to comply with the protocol requirements, fully understand the trial content, process, and possible adverse reactions, capable and willing to comply with the protocol requirements to complete this study (such as subject log recording), able to fully understand and complete the Kansas City Cardiomyopathy Questionnaire (KCCQ) questionnaire and Patient Health Questionnaire-9 (PHQ-9) scoring.

Exclusion Criteria:

1. Individuals with special clinical characteristics or disease history during screening, such as myocardial infarction, acute decompensated heart failure, hospitalization or emergency treatment due to heart failure (excluding hospitalization as specified in the trial protocol), unstable angina, stroke, or transient ischemic attack within the 30 days prior to screening or during the screening period;
2. During the screening period or on the first day of randomization, there may be laboratory tests with clinical significance, such as a 12 lead electrocardiogram indicating persistent sinus tachycardia;
3. Those who have used certain drugs or treatments before screening, such as those that may cause significant weight gain or loss within the past 3 months;
4. Based on the researcher's judgment, there are any situations that may affect the safety of the subjects or interfere with the evaluation of the trial results (such as medical, psychological, social, or geographical factors)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225 (Estimated)
Dates: Start 2025-04-10 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
The percentage change from baseline in body weight. | At week 36.

SECONDARY OUTCOMES:
The concentration of HRS-7535 in plasma. | At week 36.
The percentage change in high-sensitivity C-reactive protein (hsCRP) from baseline. | At week 36.

CONTACTS AND LOCATIONS:
Locations (1):
- Fuwai Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided